CLINICAL TRIAL: NCT02850159
Title: Effect of Simultaneous Dual Stimulation on Freezing of Gait in Parkinson's Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Yun-Hee Kim, Professor, Samsung Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2013-09-122
Record Dates: First submitted 2016-07-22; First posted 2016-07-29 (Estimated); Results first posted 2017-07-02 (Actual); Last update posted 2024-05-07 (Actual); Status verified 2024-04

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease | interventions — Transcranial Magnetic Stimulation; Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- dual-mode group (Experimental): the dual-mode NIBS with high-frequency rTMS and tDCS simultaneously
  Interventions: Device: rTMS and tDCS
- rTMS group (Active Comparator): high-frequency rTMS and sham tDCS
  Interventions: Device: rTMS

INTERVENTIONS:
Device: rTMS and tDCS — Patients underwent five consecutive daily sessions of dual-mode NIBS with high-frequency repetitive transcranial magnetic stimulation (rTMS) over the primary motor cortex of the lower leg and anodal transcranial direct current stimulation (tDCS) over the left dorsolateral prefrontal cortex simultaneously
  Arms: dual-mode group
Device: rTMS — Patients underwent five consecutive daily sessions of dual-mode NIBS with high-frequency repetitive transcranial magnetic stimulation (rTMS) over the primary motor cortex of the lower leg and sham anodal transcranial direct current stimulation (tDCS) over the left dorsolateral prefrontal cortex simultaneously
  Arms: rTMS group

SUMMARY:
The purpose of this study is to investigate the effect of dual-mode non-invasive brain stimulation (NIBS) with high-frequency repetitive transcranial magnetic stimulation (rTMS) over the primary motor cortex of the lower leg and anodal transcranial direct current stimulation (tDCS) over the left dorsolateral prefrontal cortex compared with rTMS alone in patients with Parkinson's disease (PD) with freezing of gait (FOG).

DETAILED DESCRIPTION:
Patients in the dual-mode group underwent five consecutive daily sessions of dual-mode NIBS with simultaneous high-frequency rTMS and tDCS, whereas patients in the rTMS group underwent high-frequency rTMS with sham tDCS. Assessments of FOG, motor, ambulatory and cognitive function were performed three times: at baseline before NIBS, immediately after NIBS, and one week after cessation of NIBS.

ELIGIBILITY:
Inclusion Criteria:

* diagnosed as Parkinson's disease (PD) with freezing of gait
* walk independently without walking devices

Exclusion Criteria:

* pre-existing and active major neurological diseases other than PD
* a previous history of seizures
* implanted metallic objects that would contraindicate rTMS

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2013-09; Primary Completion 2015-09 (Actual); Study Completion 2015-11 (Actual)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Chang WH, Kim MS, Park E, Cho JW, Youn J, Kim YK, Kim YH. Effect of Dual-Mode and Dual-Site Noninvasive Brain Stimulation on Freezing of Gait in Patients With Parkinson Disease. Arch Phys Med Rehabil. 2017 Jul;98(7):1283-1290. doi: 10.1016/j.apmr.2017.01.011. Epub 2017 Feb 11. PMID 28193533

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Dual-mode Group | rTMS Group
Started | 16 | 16
Completed | 16 | 16
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: 32 patients with Parkinson's disease
Groups:
- Total: Total of all reporting groups
Arm/Group | Dual-mode Group | rTMS Group | Total
Number analyzed (Participants) | 16 | 16 | 32
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.6 (7.5) | 63.8 (8.3) | 63.7 (7.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 5 | 12
  Male | 9 | 11 | 20
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 16 | 16 | 32
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Korea, Republic of | 16 | 16 | 32
Right Handedness [Count of Participants; unit: Participants] | 16 | 16 | 32

OUTCOME MEASURES:

1. Primary Outcome: Change of Freezing of Gait Questionnaire (FOG-Q)
Description: Change of a self-assessment scale for evaluating participant freezing of gait (FOG) symptoms after non-invasive brain stimulation (NIBS) for 5 consecutive days ((freezing of gait questionnaire (FOG-Q) after NIBS) - (FOG-Q before NIBS) Minimum score: -5 Maximum score: 0 Lower values represent a better outcome.
Time Frame: Assessed at T0, pre-NIBS at day 1 and T1, immediately after NIBS at day 5
Measure: Mean (Standard Deviation); unit: score
Arm/Group | Dual-mode Group | rTMS Group
Number analyzed (Participants) | 16 | 16
score | 12.0 (5.0) | 13.9 (4.9)

ADVERSE EVENTS:
Arm/Group | Dual-mode Group | rTMS Group
All-Cause Mortality (participants affected / at risk) | 0/16 | 0/16
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/16
Other Adverse Events (participants affected / at risk) | 0/16 | 0/16

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No